CLINICAL TRIAL: NCT02732730
Title: Uptake and Adherence to Daily Oral PrEP as a Primary Prevention Strategy for Young African Women: A Vanguard Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institutes of Health (NIH) (NIH); Gilead Sciences (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 082; UM1AI068619 (NIH); 12068 (Other: DAIDS)
Record Dates: First submitted 2016-03-02; First posted 2016-04-11 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: HIV
Keywords: ART (Antir-retroviral therapy); PrEP (Pre-Exposure Prophylaxis); DAIDS (Division of AIDS); HPTN (HIV Prevention Trials Network)
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Adherence Support (Experimental): For those women who choose to accept PrEP (Truvada) and assigned to receive enhanced adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Drug level counseling at Weeks 8 and 13
  Interventions: Drug: Truvada; Behavioral: Drug level counseling at Weeks 8 and 13
- Standard Adherence Support (Active Comparator): For those women who choose to accept PrEP (Truvada) and assigned to receive standard adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — 400 women who accept to initiate PrEP
  Other Names: PrEP Acceptor
Behavioral: Drug level counseling at Weeks 8 and 13 — Women who are randomized to enhanced counselling will have adherence monitoring based on plasma TFV levels obtained 4 and 8 weeks after PrEP acceptance
  Arms: Enhanced Adherence Support

SUMMARY:
To assess the acceptance rate, adherence, acceptability, and continuation of oral pre-exposure prophylaxis (PrEP) among young southern African women.

DETAILED DESCRIPTION:
A Phase IV randomized multi-site prospective study to assess PrEP acceptance and adherence among HIV-uninfected young women. All women who accept open-label daily oral PrEP will be randomized 1:1 to receive enhanced adherence counselling based on feedback from observed drug levels or standard adherence support. A subset of up to ~25 women per site (maximum 75), will participate in qualitative assessments of facilitators and barriers for PrEP acceptance, adherence and continuation.

ELIGIBILITY:
Inclusion Criteria:

Young women who meet all of the following criteria are eligible for inclusion in this study:

* Female at birth
* Age 16-25 years
* Per participant report, sexually active, defined as having vaginal or anal intercourse at least once in the month prior to screening
* Literate in one or more of the study languages
* Willing and able to provide informed consent or assent (if parental consent is required per local regulations)
* If parental consent is required per local regulations, parent/legal guardian willing and able to consent to all study procedures including HIV testing
* Able and willing to provide adequate locator information, as defined in site Standard Operating Procedures (SOPs)
* Have a score of 5 or greater on the Vaginal and Oral Intervention to Control the Epidemic (VOICE) risk score tool
* Interest in PrEP (ascertained by selected questions from the HIV Prevention Readiness Measure (HPRM) and Prep Belief Measure (PBM) defined in the Study Specific Procedures [SSP] Manual)
* Regular access to a mobile phone with SMS capacity
* Agrees not to participate in other research studies involving drugs or medical devices for the next 12 months
* Hepatitis B virus (HBV) seronegative and accepts HBV vaccination.

Exclusion Criteria:

Young women who meet any of the following criteria will be excluded from this study:

* Planning to relocate in the next 12 months
* Has a job or other obligations that would require long absences from the area (> 4 weeks at a time) for 12 months
* Any health condition that may interfere with participation, including any debilitating or life-threatening conditions
* Currently pregnant or planning to become pregnant in the next 12 months
* Any reactive or positive HIV test at Screening or Enrollment, even if subsequent testing indicates that the person is HIV-uninfected
* Renal dysfunction (Creatinine Clearance < 60 ml/min, Schwartz Equation)
* Any reported PrEP use within the last 12 months
* Concomitant participation in a clinical trial using investigational agents, including placebo-controlled clinical trials using such agents
* Prior participation in the active arm, or current participation in any arm, of an HIV vaccine trial
* Signs or symptoms of acute HIV infection (as described in the SSP Manual)
* Current active and serious infections which could interfere with study participation, including active tuberculosis infection, osteomyelitis, and all infections requiring parenteral antibiotic therapy (other than STIs requiring intramuscular injections of antibiotics); active clinically significant medical problems including poorly-controlled cardiac disease (e.g., symptoms of ischemia, congestive heart failure), or previously diagnosed malignancy expected to require further treatment.
* Current use of ARV drugs for post-exposure prophylaxis (PEP) or completion of a PEP regimen within 4 weeks prior to Screening
* History of pathological bone fracture not related to trauma
* Known allergy/sensitivity to the study drug or its components
* Receiving ongoing therapy with any of the following: investigational ARV agents, interferon or interleukin therapy, agents with substantial nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and/or other investigational agents
* Any other condition that, based on the opinion of the site Investigator of Record (IoR) or designee, would preclude provision of informed consent, make participation in the project unsafe, complicate interpretation of outcome data, or otherwise interfere with achieving the project objectives.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 451 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Study Chair — University of Washington
Locations (3):
- South Africa (2):
  - Wits Reproductive Health and HIV Institute, Johannesburg, Gauteng
  - Emavundleni CRS, Cape Town, Western Cape
- Spilhaus CRS, Harare, Belgravia, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
Data will be pooled by PID for central analysis by the Fred Hutch in Seattle, Washington

REFERENCES:
- [Derived] Magongo M, Mhlanga N, Nobanda S, Chasakara C, Yola N, Hinson K, Bryan M, Mzizi P, Essien T, Hastings N, Ndimande-Khoza MN, Bekker LG, Mgodi N, Celum C, Delany-Moretlwe S. Engagement of adolescent girls and young women into an early oral PrEP open-label study in Southern Africa: lessons learned from HPTN 082. BMC Public Health. 2025 Nov 17;25(1):3982. doi: 10.1186/s12889-025-24890-8. PMID 41249973
- [Derived] Ssemambo PK, Burton M, Mirembe BG, Nakabiito C, Donnell D, Beauchamp G, Delany-Moretlwe S, Celum C, Velloza J. Correlates of long-acting reversible contraceptive (LARC) use among young women in Southern Africa: a secondary analysis from HPTN 082. medRxiv [Preprint]. 2025 Sep 18:2025.09.16.25335943. doi: 10.1101/2025.09.16.25335943. PMID 41001449
- [Derived] Magongo M, Mhlanga N, Nobanda S, Chasakara C, Yola N, Hinson K, Bryan M, Mzizi P, Essien T, Hastings N, Ndimande-Khoza MN, Bekker LG, Mgodi N, Celum C, Delany-Moretlwe S. Recruitment of Adolescent Girls and Young Women into an Early Oral PrEP Open- Label Study in Southern Africa: Lessons Learned from HPTN 082. Res Sq [Preprint]. 2025 Mar 28:rs.3.rs-5084642. doi: 10.21203/rs.3.rs-5084642/v1. PMID 40196011
- [Derived] Beauchamp G, Hosek S, Donnell D, Chan KCG, Anderson PL, Dye BJ, Mgodi N, Bekker LG, Delany-Moretlwe S, Celum C; HPTN 082 study team. The Effect of Disclosure of PrEP Use on Adherence Among African Young Women in an Open-Label PrEP Study: Findings from HPTN 082. AIDS Behav. 2024 May;28(5):1512-1521. doi: 10.1007/s10461-023-04175-0. Epub 2023 Sep 28. PMID 37768427
- [Derived] Beauchamp G, Donnell D, Hosek S, Anderson PL, Chan KCG, Dye BJ, Mgodi N, Bekker LG, Delany-Moretlwe S, Celum C. Trust in the provider and accurate self-reported PrEP adherence among adolescent girls and young women in South Africa and Zimbabwe: HPTN 082 study. BMC Womens Health. 2023 May 19;23(1):276. doi: 10.1186/s12905-023-02418-9. PMID 37208687
- [Derived] Delany-Moretlwe S, Mgodi N, Bekker LG, Baeten JM, Li C, Donnell D, Agyei Y, Lennon D, Rose SM, Mokgatle M, Kassim S, Mukaka S, Adeyeye A, Celum C. High prevalence and incidence of gonorrhoea and chlamydia in young women eligible for HIV pre-exposure prophylaxis in South Africa and Zimbabwe: results from the HPTN 082 trial. Sex Transm Infect. 2023 Nov;99(7):433-439. doi: 10.1136/sextrans-2022-055696. Epub 2023 Mar 8. PMID 36889914
- [Derived] Beauchamp G, Hosek S, Donnell DJ, Chan KCG, Flaherty BP, Anderson PL, Dye BJ, Mgodi N, Bekker LG, Delany-Moretlwe S, Celum C; HPTN 082 study team. Development of a tool to assess HIV prevention readiness of adolescent girls and young women in HPTN 082 study. PLoS One. 2023 Feb 24;18(2):e0281728. doi: 10.1371/journal.pone.0281728. eCollection 2023. PMID 36827440
- [Derived] Velloza J, Donnell D, Hosek S, Anderson PL, Chirenje ZM, Mgodi N, Bekker LG, Marzinke MA, Delany-Moretlwe S, Celum C. Alignment of PrEP adherence with periods of HIV risk among adolescent girls and young women in South Africa and Zimbabwe: a secondary analysis of the HPTN 082 randomised controlled trial. Lancet HIV. 2022 Oct;9(10):e680-e689. doi: 10.1016/S2352-3018(22)00195-3. Epub 2022 Sep 7. PMID 36087612
- [Derived] Velloza J, Hosek S, Donnell D, Anderson PL, Chirenje M, Mgodi N, Bekker LG, Delany-Moretlwe S, Celum C; HPTN 082 study group. Assessing longitudinal patterns of depressive symptoms and the influence of symptom trajectories on HIV pre-exposure prophylaxis adherence among adolescent girls in the HPTN 082 randomized controlled trial. J Int AIDS Soc. 2021 Jun;24 Suppl 2(Suppl 2):e25731. doi: 10.1002/jia2.25731. PMID 34164929
- [Derived] Celum C, Hosek S, Tsholwana M, Kassim S, Mukaka S, Dye BJ, Pathak S, Mgodi N, Bekker LG, Donnell DJ, Wilson E, Yuha K, Anderson PL, Agyei Y, Noble H, Rose SM, Baeten JM, Fogel JM, Adeyeye A, Wiesner L, Rooney J, Delany-Moretlwe S. PrEP uptake, persistence, adherence, and effect of retrospective drug level feedback on PrEP adherence among young women in southern Africa: Results from HPTN 082, a randomized controlled trial. PLoS Med. 2021 Jun 18;18(6):e1003670. doi: 10.1371/journal.pmed.1003670. eCollection 2021 Jun. PMID 34143779
- [Derived] Velloza J, Khoza N, Scorgie F, Chitukuta M, Mutero P, Mutiti K, Mangxilana N, Nobula L, Bulterys MA, Atujuna M, Hosek S, Heffron R, Bekker LG, Mgodi N, Chirenje M, Celum C, Delany-Moretlwe S; HPTN 082 study group. The influence of HIV-related stigma on PrEP disclosure and adherence among adolescent girls and young women in HPTN 082: a qualitative study. J Int AIDS Soc. 2020 Mar;23(3):e25463. doi: 10.1002/jia2.25463. PMID 32144874

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 451 enrolled participants 427 accepted PrEP and 24 Declined. The outcomes are based on PrEP acceptors (427). Hence the total participants shown below is out of 427.
Groups:
- Standard Adherence Support: 212 women who choose to accept PrEP (Truvada) and assigned to receive standard adherence support.
- Enhanced Adherence Support: 215 women who choose to accept PrEP (Truvada) and assigned to receive enhanced adherence support.
Period: Overall Study
Arm/Group | Standard Adherence Support | Enhanced Adherence Support
Started | 212 | 215
Retention at 6 Months | 188 | 183
Completed (Patients with DBS available at 6 months) | 184 | 179
Not Completed | 28 | 36

BASELINE CHARACTERISTICS:
Groups:
- Standard Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to standard adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
- Enhanced Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to enhanced adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Drug level counseling at Weeks 8 and 13
- Total: Total of all reporting groups
Arm/Group | Standard Adherence Support | Enhanced Adherence Support | Total
Number analyzed (Participants) | 212 | 215 | 427
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [19 to 23] | 21 [19 to 22] | 21 [19 to 22]
Age, Customized [Count of Participants; unit: Participants]
  16-17 years | 11 | 16 | 27
  18-21 years | 112 | 127 | 239
  22-25 years | 89 | 72 | 161
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 215 | 427
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Zimbabwe-Shona | 70 | 66 | 136
  Zimbabwe-Ndebele | 2 | 2 | 4
  Zimbabwe-Other African Group | 1 | 4 | 5
  Zimbabwe-White | 0 | 0 | 0
  Zimbabwe-Other | 0 | 0 | 0
  South Africa-White | 0 | 0 | 0
  South Africa-Black | 139 | 143 | 282
  South Africa-Indian | 0 | 0 | 0
  South Africa-Coloured | 0 | 0 | 0
  South Africa-Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 139 | 143 | 282
  Zimbabwe | 73 | 72 | 145
Total VOICE Score [Median (Inter-Quartile Range); unit: units on a scale] — The VOICE (Validated Observational Identification of Cohort Exposure) risk scoring tool assesses HIV-1 acquisition risk using six factors scored (0-2) or (0-1), total 0-10. Higher scores indicate greater risk. Factors are (answers are worth 0 points unless otherwise noted): currently married or living with partner (if no, +2), primary partner provides financial support (if no, +1), primary partner has any other sex partner (if yes or don't know +2), past 3 months alcoholic drinks per week on average (if >1, +1), presence of STIs (if yes, +2), and age (≤25 years) (if yes, +2).
  units on a scale | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High Adherence at Six Months
Description: Number of Participants with High adherence defined as TFV-DP ≥700 fmol/punch
Time Frame: at month 6 from start of the study
Population: Among population who accepted PrEP, retained at month 6 and had detectable tenofovir diphosphate (TFV-DP) concentrations in dried blood spots (DBS)
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to receive enhanced adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Drug level counseling at Weeks 8 and 13
  * Retention at month 6
  * With DBS available
  Truvada: 400 women who accept to initiate PrEP
  Drug level counseling at Weeks 8 and 13: Women who are randomized to enhanced counselling will have adherence monitoring based on plasma TFV levels obtained 4 and 8 weeks after PrEP acceptance
- Standard Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to receive standard adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Retention at month 6
  * With DBS available Truvada: 400 women who accept to initiate PrEP
Arm/Group | Enhanced Adherence Support | Standard Adherence Support
Number analyzed (Participants) | 179 | 184
Participants | 36 | 40

2. Secondary Outcome: Number of Participants With High Adherence at Twelve Months
Description: Number of Participants with High adherence defined as TFV-DP ≥700 fmol/punch
Time Frame: 12 months from the start of the study
Population: Patients who accepted PrEP, retained at 12 months and had detectable tenofovir diphosphate (TFV-DP) concentrations in dried blood spots (DBS)
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to receive enhanced adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Drug level counseling at Weeks 8 and 13
  * Retention at month 12
  * With DBS available
  Truvada: 400 women who accept to initiate PrEP
  Drug level counseling at Weeks 8 and 13: Women who are randomized to enhanced counselling will have adherence monitoring based on plasma TFV levels obtained 4 and 8 weeks after PrEP acceptance
- Standard Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to receive standard adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Retention at month 12
  * With DBS available Truvada: 400 women who accept to initiate PrEP
Arm/Group | Enhanced Adherence Support | Standard Adherence Support
Number analyzed (Participants) | 173 | 174
Participants | 12 | 18

ADVERSE EVENTS:
Time Frame: From the start of the treatment until the resolution of all Adverse Events after completion of discontinuity of the study treatment (Up till 1 year after the start of the study treatment)
Description: For the purposes of this study, only serious adverse events (SAEs) and adverse events Grade 3 and above [with the exception of Creatinine Clearance, which will be measured using the Schwartz Equation and documented at Grade 2 or higher].
Groups:
- Standard Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to receive standard adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  Truvada: 400 women who accept to initiate PrEP
- Enhanced Adherence Support: For those women who choose to accept PrEP (Truvada) and assigned to receive enhanced adherence support, the following adherence support package will be provided:
  * Cognitive Behavioral Theory adherence support sessions
  * Two-way SMS communications
  * Optional monthly adherence support clubs
  * Drug level counseling at Weeks 8 and 13
  Truvada: 400 women who accept to initiate PrEP
  Drug level counseling at Weeks 8 and 13: Women who are randomized to enhanced counselling will have adherence monitoring based on plasma TFV levels obtained 4 and 8 weeks after PrEP acceptance
Arm/Group | Standard Adherence Support | Enhanced Adherence Support
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/215
Serious Adverse Events (participants affected / at risk) | 2/212 | 5/215
Other Adverse Events (participants affected / at risk) | 98/212 | 97/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Adherence Support (N=212) | Enhanced Adherence Support (N=215)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Adherence Support (N=212) | Enhanced Adherence Support (N=215)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 6 (7) | 5 (5)
Creatinine renal clearance decreased (Investigations) | 96 (107) | 94 (106)
Weight decreased (Investigations) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
There was very little community awareness about PrEP at the time of this study, which may have impacted adherence and persistence. We did not have the power to detect a modest effect of retrospective drug level feedback on subsequent PrEP adherence. There was not a placebo control to ethical concerns about withholding an effective intervention, so the contribution of PrEP to the low HIV incidence cannot be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT02732730/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT02732730/SAP_001.pdf